CLINICAL TRIAL: NCT03919591
Title: An Exploratory Pilot Study to Evaluate the Clinical Safety and Virologic Profile of an Experimental RSV Infection in Adults 60 to 75 Years of Age
Brief Title: RSV Study in Adults 60 to 75 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RVL-OCS-001
Record Dates: First submitted 2019-04-01; First posted 2019-04-18 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Each subject will receive one titre of the Challenge Virus intranasally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Pilot (Other): Open Label Pilot Study. All subjects will receive the viral challenge inoculum.
  Interventions: Other: Challenge virus RSV-A Memphis 37b

INTERVENTIONS:
Other: Challenge virus RSV-A Memphis 37b — Each subject will receive one titre of virus, which will be up to approximately 4.5 log10 PFU.

SUMMARY:
The purpose of this study is to infect healthy volunteers aged 60-75 years old with Respiratory Syncytial Virus (RSV) to confirm how safe and well tolerated the use of an experimental RSV virus is in a population that has not previously received the virus. Additionally, this study will also look at various components of the volunteers' blood, the lining of their noses and other samples in order to measure the effects of the virus on the body, in particularly the immune system before, during and after viral infection.

DETAILED DESCRIPTION:
RSV is a common virus that affects all human age groups. Typical RSV illness is identified by symptoms such as runny nose, stuffy nose, sneezing, sore throat, earache, malaise or tiredness, cough, shortness of breath, headache, muscle ache, joint ache or stiffness, chilliness and feverishness. RSV spreads easily from person to person through the eyes, nose or mouth when droplets containing the virus, such as those from coughing or sneezing, are inhaled or passed to others. Adults with risk factors, like another illness or disease, may experience an RSV illness that is more severe or lasts longer. RSV may also start a worsening of health in frail adults, people with weak immune systems, and those with chronic cardio-pulmonary disease.

No treatment or vaccine to treat or prevent RSV disease is available in the UK. Vaccination against RSV has the potential to be a highly beneficial and effective approach to reduce RSV disease in older adults as well as other high-risk adult and paediatric populations. The use of RSV human viral challenge model provides an important tool to evaluate the effectiveness of new RSV vaccines. Specifically, a RSV human viral challenge in 60 to 75-year-old individuals would enable measuring the effectiveness of RSV vaccines in a population that is thought to be less responsive to vaccines than the 18-45-year-old population.

The purpose of this study is to infect up to 74 healthy subjects aged 60 to 75 years old with RSV in a controlled quarantine environment to confirm how safe and well tolerated the use of an experimental RSV virus infection is in a population that has not previously received the virus. Additionally, the investigators will also look at various components of the subjects' blood, the lining of their noses and other samples in order to measure the effects of the virus on the body, in particularly the immune system before, during and after viral infection.

The study will consist of 3 phases: 1) Screening, 2) Quarantine and 3) Follow-up.

The enrolment of the subjects will be staggered with safety data reviews performed between groups. Each volunteer will be in the study for approximately 3 months from screening to their last scheduled clinic visit.

ELIGIBILITY:
Inclusion Criteria (non-exhaustive list):

* Healthy subjects aged 60 to 75 years
* Able to give informed consent
* A total body weight ≥ 50 kg and Body Mass Index (BMI) ≥ 18 kg/m2 and ≤ 33 kg/m2.
* In good health with no history of major medical conditions, or clinically significant test abnormalities that will interfere with subject safety as determined by the Investigator at screening evaluation
* Documented medical history either prior to entering the study and/or following medical history review by the Investigator at screening.
* Serum IgA result within normal range at screening.
* Subjects meeting the contraception criteria of the study.

Exclusion Criteria (non-exhaustive list):

* Subjects who have smoked ≥ 10 pack years (or 20 cigarettes a day for 10 years). Of those subjects that have smoked less than 10 pack years at any time, a subject will be excluded, if in the last year, he/she has smoked any number of cigarettes in the last month and/or they have used tobacco in any form or other nicotine-containing products in any form.
* Subjects who smoked in the last month prior to the study
* Females who are breastfeeding, have been pregnant within 6 months prior to the study, or have a positive pregnancy test.
* History of clinically significant or major disease that, in the opinion of the Investigator, may interfere with a subject completing the study and necessary investigations.
* A forced expiratory volume in 1 second (FEV1) < 80% predicted.
* Twelve-lead ECG recording with clinically relevant abnormalities.
* Positive HIV, Hep A, B or C test.
* Confirmed positive test for drugs of abuse.
* Presence of fever prior to the challenge.
* Evidence of vaccinations within the 4 weeks prior to the planned date of enrolment, or intention to receive any vaccination before the last scheduled visit of the study.
* Those employed or immediate relatives of those employed at hVIVO.
* Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior to the planned date of enrolment.
* Receipt of systemic glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of enrolment.
* History or currently active symptoms suggestive of upper or lower respiratory tract infection within 6 weeks prior to enrolment.
* Any clinically significant history of large nosebleeds.
* Any significant abnormality altering the anatomy of the nose.
* History of significant/severe wheeze, respiratory symptoms resulting in hospitalisation, or known bronchial hyperreactivity to viruses.
* History of anaphylaxis-and/or severe allergic reaction.
* Use or anticipated use during the conduct of the study of concomitant medications.
* Resident of nursing home and other long-term care facilities or with close or household contact with vulnerable people for approximately 2 weeks following discharge from unit.
* History or presence of alcohol addiction.
* Any other finding that, in the opinion of the Investigator, deems the subject unsuitable for the study.
* Subjects with no detectable antibody to the challenge virus.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Number of routine clinical assessment abnormalities reported as adverse events. | Safety data collected throughout the study (estimated 4 month).
  Multiple safety clinical parameters will be used for safety evaluation:
  * Vital signs parameters (systolic blood pressure (mmHg), diastolic blood pressure (mmHg), respiratory rate (breaths per minute), heart rate (beats per minute) and SpO2 (%)
  * Tympanic temperature (deg C)
  * Spirometry parameters (FEV1(absolute), FEV1(% predicted), Forced vital capacity (FVC) (absolute), FVC (% predicted), FEV1/FVC ratio (absolute), FEV1/FVC ratio (% predicted)
  * ECG parameters (Heart Rate (beats/min), PR interval (msec), QRS duration (msec), QT interval (msec), QTc interval (msec), QTcB interval (msec), QTcF interval (msec) and RR interval (msec))
  * Physical examination (complete examination and directed examination assessments).
Number of safety laboratory assessment abnormalities reported as adverse events. | Safety data collected throughout the study (estimated 4 month).
  * Haematology: platelet count, WBC count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, reticulocyte count, reticulocyte count [ each reported in 10^9/L]; RBC count (10^12/L), haemoglobin (g/L), haematocrit (%), MCV (fL), MCH (PG), MCHC (g/L), Haemoglobin A1c
  * Biochemistry: sodium, potassium, glucose, chloride, bicarbonate, calcium, inorganic phosphate, urea, total cholesterol [each reported in mmol/L]; uric acid, creatinine, total bilirubin, indirect bilirubin, direct bilirubin [each reported in umol/L]; serum albumin (g/L), total protein (g/L), blood urea nitrogen (mg/dL), CRP (mg/L), GGT (IU/L), ALP (IU/L), ALT (IU/L), LDH (IU/L), AST (IU/L), urea (mmol/L), total cholesterol (mmol/L), Estimated Glomerular Filtration Rate.
  * Coagulation: PT (secs), APTT (secs)
  * Cardiac Enzymes: creatine kinase (IU/L), troponin T (ng/L)
  * Urinalysis: colour, specific gravity, appearance, pH, blood, glucose, leukocytes, ketones, nitrite, protein, urobilinogen, bilirubin.
Number of subjects with study related Adverse Events (AEs) | Safety data collected throughout the study (estimated 4 month).
  * use of concomitant medications
  * frequency and severity of AEs.

SECONDARY OUTCOMES:
Viral loads/shedding measurement following inoculation with RSV | Virology and clinical data collected throughout the study (estimated 4 month).
  The AUC of RSV-A Memphis 37b viral load measured in nasopharyngeal swabs by qPCR (log10 copies/mL units) and by cell base infectivity assay (log10 copies/mL units).
Duration of viral shedding. | Virology and clinical data collected throughout the study (estimated 4 month)
  The time (in hours) from first detectable viral shedding to first undetectable viral shedding.
Measurement of the total mucus weight produced. | Virology and clinical data collected throughout the study (estimated 4 month).
  Total weight of nasal discharge (grams).
Measurement of symptoms severity by self reported symptoms diary cards. | Symptom Diary Cards data is collected throughout the quarantine period (estimated 15 days)
  Symptoms are recorded on a grading scale of 0 to 3.
Measurement of the peak tympanic temperature. | Temperature data is collected from day 0 to day 12.
  Time of the highest recorded tympanic temperature.
Number and percentage of subjects with confirmed RSV infection. | Virology data collected throughout the study (estimated 4 month)
  Confirmed infection is measured by the presence of viral shedding in nasopharyngeal swabs.
Number and percentage of subjects with Upper and Lower Respiratory Tract Infection (URTI and LRTI) | Clinical data collected throughout the study (estimated 4 month)
  URTI and LRTI are evaluated from Symptom Diary Cards and Physical Examination.

CONTACTS AND LOCATIONS:
Locations (1):
- hVIVO Services Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data might be shared with hVIVO's research partners